CLINICAL TRIAL: NCT07056647
Title: A Prospective Multicenter Randomized Controlled Trial of a Staircase Nutritional Intervention Strategy Versus Conventional ERAS Diet Management for Elderly Patients Undergoing Spinal Fusion Surgery
Brief Title: Staircase Nutritional Intervention for Elderly Patients Undergoing Spinal Fusion Surgery
Acronym: SNIEPUSFS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: xuanwu-ESN
Record Dates: First submitted 2025-06-02; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Nutritional Intervention; Spinal Surgery; Elderly; Enhanced Recovery After Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Staircase Nutritional Intervention Group (Experimental): Fourteen days before admission, different nutritional supplements will be provided according to whether the patient has diabetes and their nutritional status. Patients without diabetes who are malnourished should take enteral nutrition powder mixture three times a day, with each dose providing 265 kCal of energy. Patients without diabetes but at risk of malnutrition should take enteral nutrition powder mixture twice a day. Patients with diabetes who are malnourished should take low - sugar whole - protein enteral nutrition powder three times a day, with each dose providing 250 kCal of energy. Patients with diabetes and at risk of malnutrition should take low - sugar whole - protein enteral nutrition powder twice a day.
  During the peri - operative period, a strict 6 - hour fasting of solid food and 2 - hour fasting of clear liquid before surgery is implemented. Two hours after surgery, all patients should take multi - dimensional carbohydrates, which provide 115 kCal of energy. Four h
  Interventions: Dietary Supplement: Staircase Nutritional Intervention
- Standard ERAS Diet Management Group (Active Comparator): Only nutritional education is provided to patients before admission, without any specific nutritional supplements. During the peri - operative period, patients are required to fast from food and water for 8 hours before surgery. Six hours after surgery, patients are allowed to drink water. They can start consuming liquid food after passing gas from the anus. No specific energy - containing nutritional supplements are given during this period. A nutritional guidance manual is distributed to patients upon discharge, and there are no targeted nutritional interventions or follow - up measures related to energy intake subsequently.
  Interventions: Dietary Supplement: Standard ERAS Diet Management Group

INTERVENTIONS:
Dietary Supplement: Staircase Nutritional Intervention — Fourteen days before admission, different nutritional supplements will be provided according to whether the patient has diabetes and their nutritional status. Patients without diabetes who are malnourished should take enteral nutrition powder mixture three times a day, with each dose providing 265 kCal of energy. Patients without diabetes but at risk of malnutrition should take enteral nutrition powder mixture twice a day. Patients with diabetes who are malnourished should take low - sugar whole - protein enteral nutrition powder three times a day, with each dose providing 250 kCal of energy. Patients with diabetes and at risk of malnutrition should take low - sugar whole - protein enteral nutrition powder twice a day.
  During the peri - operative period, a strict 6 - hour fasting of solid food and 2 - hour fasting of clear liquid before surgery is implemented. Two hours after surgery, all patients should take multi - dimensional carbohydrates, which provide 115 kCal of energy. Four ho
  Arms: Staircase Nutritional Intervention Group
Dietary Supplement: Standard ERAS Diet Management Group — Only nutritional education is provided to patients before admission, without any specific nutritional supplements. During the peri - operative period, patients are required to fast from food and water for 8 hours before surgery. Six hours after surgery, patients are allowed to drink water. They can start consuming liquid food after passing gas from the anus. No specific energy - containing nutritional supplements are given during this period. A nutritional guidance manual is distributed to patients upon discharge, and there are no targeted nutritional interventions or follow - up measures related to energy intake subsequently.
  Arms: Standard ERAS Diet Management Group

SUMMARY:
The goal of this prospective multicenter randomized controlled clinical trial is to evaluate the efficacy of a staircase nutritional intervention in reducing postoperative complications and improving long-term functional recovery in elderly patients aged ≥75 years scheduled for spinal fusion surgery. The main questions it aims to answer are:

1. Does the staircase nutritional intervention reduce the 30-day postoperative complication rate, as measured by the Comprehensive Complication Index (CCI), compared to conventional ERAS diet management?
2. Does the staircase nutritional intervention improve 1-year functional recovery, as assessed by Oswestry/Neck Disability Index (ODI/NDI) and health-related quality of life (EQ-5D), compared to conventional ERAS diet management?

Researchers will compare the intervention group receiving MNA - based staircase nutritional intervention (including 14-day preadmission oral nutritional supplementation, perioperative personalized nutritional support, and postdischarge continuous management) combined with surgery-specific prehabilitation training to the control group receiving conventional ERAS diet management to see if the former leads to better clinical outcomes and long-term functional recovery.

Participants will

Undergo randomization: Be randomly assigned to either the intervention group or the control group.

Receive assigned interventions:

Control group: Receive conventional ERAS diet management, including preadmission nutritional education and early postoperative oral intake.

Intervention group: Undergo MNA - based staircase nutritional intervention and surgery-specific prehabilitation training.

Participate in follow-up: Complete short-term (within 90 days postoperatively) and long-term (6 and 12 months postoperatively) follow-up assessments, including laboratory tests, functional evaluations, and satisfaction surveys.

DETAILED DESCRIPTION:
Lumbar degenerative diseases are one of the common conditions in the elderly population, primarily characterized by pain and functional decline in the affected area, often accompanied by poorer health-related quality of life (HRQoL). Studies predict that by 2025, the global population aged 75 and over will double compared to 2019, exceeding 1.5 billion, and the number of patients with degenerative spinal diseases will increase accordingly, imposing a huge economic burden on healthcare systems. For elderly patients with degenerative spinal diseases who fail conservative treatment, surgical decompression and fusion remains a key measure to alleviate clinical symptoms and improve long-term prognosis. However, up to 40% of hospitalized elderly patients suffer from malnutrition. Many studies have confirmed that malnourished surgical patients have higher rates of postoperative mortality, morbidity, longer hospital stays, readmission rates, and hospitalization costs.

In response to the adverse effects of malnutrition in the elderly population, spinal surgery clinics have made efforts to address this issue. Enhanced Recovery After Surgery (ERAS) is a multidisciplinary collaborative care model based on evidence-based medicine, which optimizes a series of perioperative (preoperative, intraoperative, postoperative) management measures to reduce surgical stress responses, lower complication rates, accelerate patient recovery, and shorten hospital stays. Its core lies in improving traditional perioperative management processes by integrating the latest research achievements from multiple disciplines, including nutrition. Spinal surgery introduced ERAS into perioperative processes more than a decade ago. Through continuous application and updates, ERAS has provided important guarantees for perioperative nutritional management in spinal surgery. By delivering short-term nutritional support and early postoperative oral intake strategies, it effectively promotes postoperative gastrointestinal recovery, improves patient satisfaction, and, in conjunction with other ERAS components, reduces infection-related complications and shortens hospital stays. However, the nutrition-related management in perioperative enhanced recovery is not a strict nutritional intervention, and its impact on improving patients' nutritional status is limited. Therefore, implementing longer-term perioperative nutritional interventions for malnourished patients is of practical significance. Guidelines indicate that oral nutritional supplements (ONS) are an effective form of nutritional intervention for patients. Before nutritional intervention, nutritional risk assessment is required. The Mini-Nutritional Assessment (MNA), a nutritional screening tool specifically developed for elderly patients, has been adopted in many studies to guide nutritional interventions, and its effectiveness has been fully validated. MNA can effectively stratify patients by evaluating 18 items, including dietary intake, weight changes, mobility, and disease status, classifying nutritional status into three tiers: well-nourished (>24 points), at risk of malnutrition (17-23.5 points), and malnourished (<17 points). Oral nutritional supplements (ONS), available in liquid, powder, or paste forms, offer advantages of convenient oral administration and physiological absorption, making them highly suitable for elderly patients with reduced appetite, eating ability, and gastrointestinal capacity. Numerous studies have confirmed that ONS can effectively improve serum protein levels in malnourished patients, reduce the risk of postoperative complications, and accelerate recovery. Historically, the diagnosis and treatment of spinal degenerative diseases have always centered on surgery. However, surgical trauma represents a significant event that accelerates aging in elderly patients. Many patients who have suffered from spinal degenerative diseases for years often forgo surgical opportunities due to perceived high potential risks, continuing to endure pain. In recent years, the concept of prehabilitation has brought hope to elderly patients. When facing fusion surgery, elderly patients are not merely passive bearers of risks. Unlike non-modifiable preoperative factors such as age and comorbidities, nutritional reserve- a key characteristic of elderly patients-is considered improvable. Based on previous research experience, preoperative nutritional interventions to enhance the nutritional status of elderly patients can help reduce postoperative complications, accelerate postoperative recovery, and potentially yield long-term benefits. Current related research has significant limitations: few studies focus on nutritional interventions for patients undergoing spinal fusion surgery; the limited clinical studies in relevant populations are confined to short-term in-hospital interventions and outcomes; and intervention protocols lack stage-specific design. These shortcomings severely restrict the generalizability of perioperative nutritional intervention protocols for elderly spinal surgery patients.

Research Objective This study aims to conduct a prospective multicenter randomized controlled trial enrolling elderly patients aged ≥75 years scheduled for spinal fusion surgery. Using nutritional stratification, it will compare a staircase nutritional intervention with conventional ERAS diet management, evaluating 30-day postoperative complication rates and 1-year functional recovery outcomes. The goal is to establish an optimized perioperative nutritional protocol for elderly spinal fusion patients, filling the research gap in long-term stage-specific interventions and improving surgical safety and long-term quality of life for this population.

Study Design and Implementation This is a prospective, multicenter, parallel-group randomized controlled trial conducted across multiple teaching hospitals. Control group patients will receive conventional ERAS diet management, including preadmission nutritional education and early postoperative oral intake. The intervention group will undergo MNA-based staircase nutritional interventions, covering 14-day preadmission oral nutritional supplementation (ONS), perioperative personalized nutritional support, and postdischarge continuous management, combined with surgery-specific prehabilitation training. The study will commence in July 2025, with a 12-month enrollment period and a 12-month follow-up period. The total study duration is 30 months, with data collection and analysis expected to be completed by January 2028.

Primary Outcome The primary outcome is the Comprehensive Complication Index (CCI), a continuous scale (0-100 points, where 100 indicates death due to complications) that integrates all complications and their severity based on the Clavien-Dindo classification system. Postoperative complications will be recorded up to 90 days post-surgery (definitions in Appendix 1), with severity scored using the Clavien-Dindo system. CCI will be calculated using an online calculator (http://www.assessurgery.com). Previous studies have validated CCI as an effective measure of postoperative morbidity, demonstrating greater comprehensiveness and sensitivity than traditional metrics (e.g., overall complication rate or severe complication rate) for surgical research endpoints.

Secondary Outcomes

Pain level and pain-related functional limitation: Assessed using the Visual Analogue Scale (VAS) and Oswestry/Neck Disability Index (ODI/NDI).

Physiological function recovery: Sum of days to first defecation, first urination, and first ambulation postoperatively.

Laboratory indicators: Serum albumin, hemoglobin, Prognostic Nutritional Index (PNI), and inflammatory markers (C-reactive protein [CRP]) monitored on postoperative days 1, 3, and pre-discharge.

Health-related quality of life: Evaluated using the EuroQol five-dimension scale (EQ-5D, 0 = poorest health, 100 = best health).

Physical function: Assessed via 6-meter walking speed and handgrip strength. Patient satisfaction: Measured using the North American Spine Society (NASS) satisfaction scale (1-4 points, where 1 = most satisfied, 4 = least satisfied), with responses categorized as: treatment met expectations (1 point); improvement below expectations but willing to undergo the same treatment (2 points); improvement below expectations and unwilling to undergo the same treatment (3 points); same or worse than preoperative status (4 points).

Discharge Criteria

1. Complete or major resolution of preoperative symptoms, or treatment meets the patient's expectations;
2. No surgical-related complications, or complications are controlled;
3. No further need for clinical treatment.

Follow-Up Indicators

Short-term follow-up (within 90 days postoperatively): Record primary and total hospital stay durations, non-home discharge rate, readmission rate, unplanned readmission data within 90 days, and postoperative outcomes.

Long-term follow-up (6 and 12 months postoperatively):

Function and quality of life:

Pain level: Visual Analogue Scale (VAS). Functional disability: Oswestry Disability Index (ODI, for lumbar patients), Neck Disability Index (NDI, for cervical patients).

Activities of daily living: ADL and Instrumental Activities of Daily Living (IADL) scales.

Quality of life: EQ-5D score.

Clinical and imaging evaluations:

Readmission rate: Frequency and causes of readmission due to surgery-related complications (e.g., infection, internal fixation issues).

Imaging fusion rate (lumbar/thoracolumbar fusion patients): Assessment of surgical segment bone fusion via X-ray or CT (success defined as continuous bony bridge formation).

Long-term complications: Incidence of internal fixation failure, adjacent segment degeneration, chronic pain, etc.

Long-term nutritional status: Serum albumin and hemoglobin levels at 1 year postoperatively to assess malnutrition recurrence risk.

ELIGIBILITY:
Inclusion Criteria:

* Age and Gender: Aged ≥ 75 years, regardless of gender. Surgery Type: Scheduled for elective spinal fusion surgery, including but not limited to lumbar, thoracic, and cervical spinal fusion surgeries. The surgeries are aimed at treating spinal degenerative diseases (such as lumbar disc herniation, lumbar spinal stenosis, etc.), spinal trauma, spinal deformities, etc.

Nutritional Status: Willing and able to cooperate with nutritional assessments (such as Mini - Nutritional Assessment, MNA), and patients with any level of nutritional risk are included.

Physical Condition: American Society of Anesthesiologists (ASA) physical status classification Ⅰ - Ⅲ, meaning the physical condition is relatively tolerable for surgery, without severe failure of important organs such as the heart, lungs, liver, and kidneys, and without uncontrolled severe hypertension, diabetic ketoacidosis, and other acute complications.

Cognitive and Communication Ability: Possessing basic cognitive and communication abilities, being able to understand the purpose, process, and relevant requirements of the study, and signing a written informed consent form.

Life Expectancy: With a life expectancy of more than 1 year to facilitate long - term postoperative follow - up and assessment.

Exclusion Criteria:

* Severe Underlying Diseases: Presence of severe heart failure (New York Heart Association functional class Ⅳ), end - stage liver disease (such as decompensated liver cirrhosis with severe ascites, hepatic encephalopathy, etc.), end - stage renal disease (requiring maintenance dialysis treatment), end - stage malignant tumors, and other serious underlying diseases that severely affect life and health and recovery.

Psychiatric and Neurological Diseases: Suffering from severe mental illnesses (such as schizophrenia, major depressive disorder in the acute phase and unable to cooperate with the study), Alzheimer's disease and unable to understand the content of the study, and serious neurological diseases (such as long - term bedridden patients with severe stroke and impaired consciousness).

Contraindications to Nutritional Supplements: Allergic to the components of the nutritional supplements involved in the study (such as enteral nutrition powder mixture, low - sugar whole - protein enteral nutrition powder, etc.) or having severe intolerance.

Recent Special Situations: Having a history of severe trauma or major surgery (other than the planned spinal fusion surgery) in the past 3 months; having a history of severe gastrointestinal diseases such as gastrointestinal bleeding and intestinal obstruction in the past 1 month.

Others: Currently participating in other clinical trials that may affect the results of this study; having insurmountable compliance problems (such as failure to take nutritional supplements on time, refusal of follow - up, etc.).

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Comprehensive Complication Index (CCI) | up to 90 days after surgery
  The primary outcome is the Comprehensive Complication Index (CCI), a continuous scale (0-100 points, where 100 indicates death due to complications) that integrates all complications and their severity based on the Clavien-Dindo classification system. Postoperative complications will be recorded up to 90 days post-surgery (definitions in Appendix 1), with severity scored using the Clavien-Dindo system. CCI will be calculated using an online calculator (http://www.assessurgery.com). Previous studies have validated CCI as an effective measure of postoperative morbidity, demonstrating greater comprehensiveness and sensitivity than traditional metrics (e.g., overall complication rate or severe complication rate) for surgical research endpoints.

SECONDARY OUTCOMES:
Pain level | up to 90 days after surgery
  The Visual Analogue Scale (VAS) is a widely used tool to measure pain intensity. It consists of a 10-centimeter horizontal line, with endpoints labeled "no pain" (0) and "worst possible pain" (10). During the assessment, patients are asked to mark a point on the line that corresponds to their current pain level. This simple yet effective method provides a quantitative measure of pain, allowing for consistent monitoring and comparison of pain intensity over time.
Physiological function recovery | up to 90 days after surgery
  Sum of days to first defecation, first urination, and first ambulation postoperatively.
Serum Albumin Levels Measured Postoperatively | up to 90 days after surgery
  Serum albumin is a protein produced by the liver and is an important marker of nutritional status and overall health. To measure serum albumin levels, a blood sample is drawn and analyzed in a clinical laboratory using techniques such as spectrophotometry. Normal serum albumin levels typically range from 3.5 to 5.0 grams per deciliter (g/dL). In the postoperative period, monitoring serum albumin helps assess a patient's recovery, as low levels may indicate poor nutrition, inflammation, or other complications that can delay healing.
Health-related quality of life | up to 90 days after surgery
  Evaluated using the EuroQol five-dimension scale (EQ-5D, 0 = poorest health, 100 = best health).
Physical function | up to 90 days after surgery
  Assessed via 6-meter walking speed and handgrip strength.
Patient satisfaction | up to 90 days after surgery
  Measured using the North American Spine Society (NASS) satisfaction scale (1-4 points, where 1 = most satisfied, 4 = least satisfied), with responses categorized as: treatment met expectations (1 point); improvement below expectatio
Functional Disability Assessment Using Oswestry/Neck Disability Index (ODI/NDI) | up to 90 days after surgery
  The Oswestry Disability Index (ODI) and Neck Disability Index (NDI) are self-report questionnaires designed to evaluate the functional disability caused by low back pain (ODI) or neck pain (NDI), respectively. Each index contains a series of questions related to daily activities such as personal care, lifting, walking, and sleeping. Patients rate their difficulty performing these activities on a scale from 0 (no disability) to 5 (complete disability). The total score is calculated as a percentage, with higher scores indicating greater disability. These indices are crucial for assessing the impact of spinal conditions on a patient's quality of life and tracking the effectiveness of treatments.
Hemoglobin Concentrations in Postoperative Blood Samples | up to 90 days after surgery
  Hemoglobin is a protein in red blood cells responsible for carrying oxygen throughout the body. Hemoglobin levels are measured by taking a blood sample, which is then analyzed to determine the amount of hemoglobin present, usually expressed in grams per deciliter (g/dL). Normal hemoglobin levels vary by age and gender, with typical ranges being 13.5-17.5 g/dL for adult males and 12.0-15.5 g/dL for adult females. Postoperatively, monitoring hemoglobin is essential to detect blood loss, anemia, or other conditions that may affect oxygen delivery to tissues and overall recovery.
Calculation of Prognostic Nutritional Index (PNI) Postoperatively | up to 90 days after surgery
  The Prognostic Nutritional Index (PNI) is a composite score used to predict the risk of postoperative complications and overall prognosis based on a patient's nutritional and inflammatory status. It is calculated using the following formula: PNI = 10 × serum albumin (g/dL) + 0.005 × total lymphocyte count (/mm³). A higher PNI generally indicates better nutritional status and a lower risk of complications, while a lower score suggests increased vulnerability. PNI is calculated using blood test results obtained on postoperative days 1, 3, and pre-discharge to guide clinical decision-making and optimize patient care.
C-reactive Protein (CRP) Levels as an Inflammatory Marker Postoperatively | up to 90 days after surgery
  C-reactive protein (CRP) is an acute-phase protein produced by the liver in response to inflammation, infection, or tissue injury. CRP levels are measured by analyzing a blood sample in a laboratory, typically using immunoassay techniques, and are expressed in milligrams per liter (mg/L). Normal CRP levels are usually less than 5 mg/L. Elevated CRP levels postoperatively can indicate the presence of inflammation, such as an infection at the surgical site or a systemic response to tissue damage. Monitoring CRP on postoperative days 1, 3, and pre-discharge helps healthcare providers assess the healing process and detect potential complications early.

OTHER OUTCOMES:
Long-term follow-up of Postoperative Pain Level Measured by Visual Analogue Scale (VAS) | 6 and 12 months postoperatively
  The pain level is evaluated using the Visual Analogue Scale (VAS), a 10-centimeter horizontal line with endpoints labeled "no pain" (0) and "worst possible pain" (10). Patients mark a point corresponding to their current pain intensity at follow-up visits, quantifying pain to monitor changes over time.
Long-term follow-up of functional disability assessment using Oswestry/NDI Index | 6 and 12 months postoperatively
  Functional disability is assessed with the Oswestry Disability Index (ODI) for lumbar patients and Neck Disability Index (NDI) for cervical patients. Self-report questionnaires include daily activities (e.g., personal care, walking), rated 0 (no disability) to 5 (complete disability). Total scores (as percentages) reflect disability severity and treatment impact.
Long-term follow-up of ADL and IADL scales assessment of activities of daily living | 6 and 12 months postoperatively
  ADL (basic self-care: eating, dressing) and IADL (complex skills: shopping, finance) scales evaluate independent living abilities. Scores at follow-up visits determine recovery and surgical impact on daily function.
Long-term follow-up of quality of life evaluation by EQ-5D score | 6 and 12 months postoperatively
  The EQ-5D scale assesses mobility, self-care, pain, and mental state (5 dimensions, each 0-3 severity levels). A visual analog health rating (0-100) is integrated to generate scores, with higher values indicating better quality of life.
Long-term follow-up of readmission rate and associated causes due to surgery-related complications | 6 and 12 months postoperatively
  Readmissions within follow-up periods for complications (infection, internal fixation issues) are counted, with causes analyzed to assess surgical safety and long-term risks.
Long-term follow-up of imaging fusion rate assessment of surgical segment in lumbar/thoracolumbar fusion patients | 6 and 12 months postoperatively
  X-ray/CT evaluates bony fusion at the surgical segment, defined by continuous bony bridge formation. Fusion rates are calculated to monitor healing and surgical outcomes.
Long-term follow-up of incidence of long-term complications | 6 and 12 months postoperatively
  Complications (internal fixation failure, adjacent segment degeneration, chronic pain) are tracked to evaluate long-term surgical impact and patient prognosis.
Long-term follow-up of long-term nutritional status assessment by serum albumin and hemoglobin levels | 6 and 12 months postoperatively
  Serum albumin (3.5-5.0 g/dL normal) and hemoglobin (13.5-17.5 g/dL for males, 12.0-15.5 g/dL for females) are measured at 1-year follow-up to assess malnutrition risk and long-term health.

CONTACTS AND LOCATIONS:
Overall Officials: Shibao Lu, MD, Study Chair — Xuanwu Hospital of Capital Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Millrose M, Schmidt W, Krickl J, Ittermann T, Ruether J, Bail HJ, Gesslein M. Influence of Malnutrition on Outcome after Hip Fractures in Older Patients. J Pers Med. 2023 Jan 3;13(1):109. doi: 10.3390/jpm13010109. PMID 36675770
- [Result] Yap YY, Tan SH, Choon SW. Elderly's intention to use technologies: A systematic literature review. Heliyon. 2022 Jan 13;8(1):e08765. doi: 10.1016/j.heliyon.2022.e08765. eCollection 2022 Jan. PMID 35128090